CLINICAL TRIAL: NCT03373357
Title: Hypertension and Cardiovascular Risk Associated With Obstructive Sleep Apnea in Adult in Guadeloupe (French West Indies)
Acronym: HTA-SAHOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RBM-PAP- 2007/19
Record Dates: First submitted 2017-12-04; First posted 2017-12-14 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Hypertension Arterial
Keywords: sleep apnea; arterial hypertension; cardiovascular risk
MeSH Terms: conditions — Hypertension; Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: All the patients will have sampling blood specific to the protocol:
  * Insulinémie
  * US CRP(TEACHERS' CENTRE)
  * Implementation of a sérothèque
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient not SAHOS (Other): The medical follow-up of patients no SAHOS will be assured by the investigators of the unity of cardiovascular explorations: phone consultation in 1 month, 3mois, then every 6 months, and an annual visit.
  Interventions: Other: Patient not SAHOS
- Patient SAHOS sailed by the ventilation in PPC and not sailed (Other): The patients who have a SAHOS sailed by the ventilation in PPC will be estimated and followed in 3 months then every 6 months by the investigators of the service of pneumology and the unity of cardiovascular explorations. The control of the material and its tolerance, the data supplied by the service providers (bodies of ventilation at home) will be estimated by the investigator of the service of pneumology. IDE the unity of cardiovascular explorations will plan and will realize a 2nd one MAPA after 3 months of ventilation in PPC.
  Interventions: Other: Patient SAHOS sailed by the ventilation in PPC and not sailed

INTERVENTIONS:
Other: Patient not SAHOS — Phone consultation in 1 month, 3mois, then every 6 months, and an annual visit.
  * Cardiovascular events arisen during the duration of the study
  * Modifications of the lifestyle: alcohol, physical activity
  * Weight
  * Clinical measure of the PA
  * Clinical examination
  * The collection of the cardiovascular events arisen during the duration of the study will be realized for all the inclusive patients
  Arms: Patient not SAHOS
Other: Patient SAHOS sailed by the ventilation in PPC and not sailed — Questionnaire of subjective evaluation of diurnal slumber: scale of Epworth and search for appearance of at least 2 of the following symptoms: sleep not salvage dealer, night-breathlessnesses, multiple awakenings, fatigue, disordersconfusions, nycturie, snore.
  * Questionnaire of evaluation of the global quality of life of the SAHOS
  * Appearance of new cardiovascular risk factors
  * Cardiovascular events arisen during the duration of the study
  * Modification of the current treatments
  * Modifications of the lifestyle: alcohol, physical activity
  * Weight
  * Clinical measure of the PA
  * Clinical examination
  * The collection of the cardiovascular events arisen during the duration of the study will be realized for all the inclusive patients
  Arms: Patient SAHOS sailed by the ventilation in PPC and not sailed

SUMMARY:
The MAPA is the reference method to estimate the PA during the SAHOS. The MAPA can be recommended over 48 hours: indeed, the PA falls at the beginning of every apnea then increases gradually up to a pressif peak arising at the time of the ventilatoire resumption. These variations arise under the influence of 4 stimulus: the désaturation in O2, the rise of the PaCO2, the increase of the respiratory effort and the microawakening of the end of apnea who are at the origin of a sympathetic stimulation.

Consequently a better diagnostic approach of the HTA (confirmation of a resistant HTA, an identification of the masked HTA and the patients " not dipper " by the MAPA), the identification of the SAHOS, and a better coverage) of the associated cardiovascular risk factors are essential and establish a stake in public health.

To investigator's knowledge, no datum or study on the association HTA-SAHOS and its consequences was until then realized in the French overseas departments.

DETAILED DESCRIPTION:
In Guadeloupe, data on the relationships between arterial hypertension and obstructive sleep apnea are unavailable. The aim of this study was: to assess the frequency of hypertension and non-dipper pattern evaluated by 48-hour ambulatory blood pressure monitoring in an adult population identified obstructive sleep apnea/non-obstructive sleep apnea during overnight polygraphy ; to determine the cardio-metabolic factors associated with obstructive sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* Patient suspected of SAHOS;
* Patient or third-party responsible for receiving information on the study and who signed informed consent ;
* Patient age over 18 years; Patient living in Guadeloupe.

Exclusion Criteria:

* Patient non-affiliated to the social security scheme ;
* Patient with obstructive bronchopneumopathy, neuro-muscular pathology,
* central and mixed SAS, cardiac arrhythmia,
* systemic and chronic inflammatory syndrome ; -
* Pregnant and lactating patient ;
* patient in emergency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2008-09-09 (Actual); Primary Completion 2014-11-19 (Actual); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
the frequency of hypertension | At the of the enrollment period, an average of 3 years", etc.).
  The primary outcome measure the frequency of hypertension and non-dipper pattern evaluated by 48-hour ambulatory blood pressure monitoring in an adult population identified obstructive sleep apnea/non-obstructive sleep apnea during overnight polygraphy.

SECONDARY OUTCOMES:
The cardio-metabolic factors | "through study completion, an average of 8 years"
  All the enrolled patients will be followed during 5 years and particularly concerning:
  * the appearance of new risk cardiovascular factors
  * the advent of cardiovascular events

CONTACTS AND LOCATIONS:
Overall Officials: Rachel BILLY BRISSAC, Dorctor cardiovascular, Principal Investigator — Hospital University Center of Pointe-à-Pitre
Locations (1):
- Hospital University Center of Pointe-à-Pitre, Pointe-à-Pitre, Guadeloupe

IPD SHARING:
Plan to Share IPD: No